CLINICAL TRIAL: NCT00071370
Title: Activating Effects of Sleep Deprivation On Synchronized MEG-EEG Recordings Of Epilepsy Patients With Non-Diagnostic EEG
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040015; 04-N-0015
Record Dates: First submitted 2003-10-20; First posted 2003-10-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Epilepsy
Keywords: Magnetoencephalography; Electroencephalogram (EEG); Interictal Epileptiform Discharges; Epilepsy; Sleep Deprivation; Seizure
MeSH Terms: conditions — Epilepsy; Sleep Deprivation; Seizures

SUMMARY:
This study will evaluate how the state of being completely deprived of sleep has an effect on recordings of magnetoencephalography (MEG) and electroencephalography (EEG), in relation to how alert someone is and how sleepy someone perceives himself or herself to be. EEG measures electronic potential differences on the scalp. On the other hand, MEG is a non-invasive technique for recording the activity of neurons in the brain, through recording of magnetic fields caused by synchronized neural currents. It has the ability to detect seizures. Because magnetic signals of the brain vary, this technique must balance two key problems: weakness of the signal and strength of the noise. The EEG is sensitive to extra-cellular volume currents, whereas the MEG primarily registers intra-cellular currents. Because electrical fields are quite dependent on the conductive properties of the tissues, and magnetic fields are significantly less distorted by tissue, the MEG has better spatial resolution. There is a great deal of evidence that EEG and MEG provide complementary data about underlying currents of ions.

The complex relationship of sleep and epilepsy is well known. Sleep has been used for many years as a powerful EEG activator. Many researchers have supported the hypothesis that there is a specific activating effect of sleep deprivation on epileptic discharges. Sleep deprivation is defined as a sleepless state of longer than 24 hours. The increased use of MEG in diagnosis could improve the procedure for evaluating patients before surgery for epilepsy, by making invasive studies less necessary.

Patients 18 years of age or older, with a diagnosis of epilepsy and with a documented last routine EEG (at least 2 weeks earlier) and routine EEG on the day of a baseline MEG-EEG without interictal epileptiform discharges (IEDs) may be eligible for this study.

Participants will be rated according to the Epworth, Stanford, and Karolinska Sleepiness Scales, to determine their subjective sleepiness. They will be randomly assigned to stay awake all night or sleep in the hospital overnight. That is, a sleep deprivation and non-sleep deprivation synchronized MEG-EEG recording will be performed in random order. Then the sequence of sleep deprivation and non-sleep deprivation will be reversed within 14 to 21 days. During the recordings, the patient will either sit or lie with his or her head in a helmet covering the entire head, with openings for the eyes and ears. Brain magnetic fields will be recorded with a 275-channel OMEGA system. Throughout the session, visual and two-way audio communication will be maintained with the patient. Recording sessions will last 90 to 180 minutes, with the patient allowed to take breaks after at least 10 minutes in a scanner. Attempts will be made to encourage patients to stay awake and sleep for about the same amount of time during each recording, to acquire comparable amounts of sleep and awake recordings.

DETAILED DESCRIPTION:
Objective:

We would like to evaluate the activating effects of complete sleep deprivation (SD) on synchronized MEG-EEG recordings, and on each of the components singly, in relation to the degree of alertness during recording (awake vs. sleep) and the subjective degree of sleepiness as assessed by standardized scales. We postulate that acute SD will increase the diagnostic yield of synchronized MEG-EEG and activate both modalities (MEG, EEG) to the same degree. The increased diagnostic utility of MEG could improve the epilepsy surgery evaluation procedure for many patients by rendering invasive studies less necessary. The medical and economic utilization of such expensive resources as MEG could thus be rationalized.

Population:

Participants of this study will be epilepsy patients whose last routine interictal EEG (performed at least two weeks earlier), subsequent pre-screening EEG and screening MEG-EEG show no interictal epileptiform discharges (IEDs), and are therefore considered non-diagnostic.

Study Design/Methods:

We will use a 275-channel Whole-head MEG System (CTF Systems 2001 Inc.). Patients will have a screening, non-SD and SD MEG-EEG after their degree of sleepiness is assessed using the Epworth, Stanford and Karnolinska sleepiness scales. Starting one day after the MEG-EEG, SD and non-SDMEG-EEG will be performed in random order within 14-21 days of each other. This will ensure an equal amount of sampling effect in SD and non-SD data sets. The MEG-EEG session will last 90 to 180 minutes. Patients may take a break after at least 10 minutes in a scanner. We will attempt to record a comparable amount of awake and sleep data. At least thirty minutes of artifact-free baseline, non-SD and SD MEG-EEG will be analyzed. For the purpose of blinding, each modality will be read independently by two readers, each of whom will be blinded to the relationship of the MEG-EEG data to sleep deprivation, results obtained by the other modality and subjective degree of sleepiness. Only interpretations of each modality agreed upon by both readers will be accepted. When there is no agreement, a third independent reader will resolve the disagreement.

Outcomes:

The primary outcome measure will be the proportion of seizure foci detected and delineated after SD on synchronized MEG-EEG recordings. Comparisons will also be made for each recording modality and between them, according to the state of alertness during recording and subjective feeling of sleepiness before each recording.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients 18 years or older

Patients of both sexes and of any race or ethnicity who have a diagnosis of epilepsy routine EEG on the day of a baseline MEG-EEG without IEDs.

EXCLUSION CRITERIA:

Patients younger than 18 years

Patients with progressive neurological disorders

Patients who are unable to lie still or cooperate adequately with MRI or MEG/EEG

Patients who are unable to sustain the required degree of sleep deprivation.

Patients who have had brain surgery.

Patients unable to sign and understand the study consent

Patients with IEDs on a routine EEG

Patients with IEDs on the baseline MEG-EEG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2003-10; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dinner DS. Effect of sleep on epilepsy. J Clin Neurophysiol. 2002 Dec;19(6):504-13. doi: 10.1097/00004691-200212000-00003. PMID 12488781
- [Background] Brockhaus A, Lehnertz K, Wienbruch C, Kowalik A, Burr W, Elbert T, Hoke M, Elger CE. Possibilities and limitations of magnetic source imaging of methohexital-induced epileptiform patterns in temporal lobe epilepsy patients. Electroencephalogr Clin Neurophysiol. 1997 May;102(5):423-36. doi: 10.1016/s0921-884x(97)96625-x. PMID 9191586
- [Background] el-Ad B, Neufeld MY, Korczyn AD. Should sleep EEG record always be performed after sleep deprivation? Electroencephalogr Clin Neurophysiol. 1994 Apr;90(4):313-5. doi: 10.1016/0013-4694(94)90150-3. PMID 7512913